CLINICAL TRIAL: NCT01661062
Title: A Pilot Study of Tumor and Critical Normal Tissue Motion in Head and Neck Cancer Using Cone Beam CT
Brief Title: A Study Using Cone Beam CT for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005.084; HUM 757 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2011-09-26; First posted 2012-08-09 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cone Beam CT (Experimental): All patients will be included in the treatment arm of this study. For the purposes of this study patients will get CT scans every day for the length of their radiation therapy (in order to assess if CT every day provides additional information compared with CT scans performed less frequently). Although the exact amount of radiation patients get will be determined by their doctor, it is expected that they will get approximately 7 weeks, approximately 35 total cone beam CT scans.
  Interventions: Other: Cone Beam Computed Tomography (CT) Scan

INTERVENTIONS:
Other: Cone Beam Computed Tomography (CT) Scan — Cone beam CT scan is considered a noninvasive procedure (meaning that the procedure does not require breaking the skin or any tools that physically enter the body). It will add a small amount of additional radiation dose (less than 1%) to the head and neck. The increase in the amount of radiation is only a very small amount more than what patients who get standard daily imaging receive. The amount of radiation from the cone beam CT scans is not significant (less than 1%) when compared to the amount of radiation generally received for treatment of head and neck cancer.
  Other Names: CBCT

SUMMARY:
Cone beam CT (computed tomography) is a developing technology which allows CT images to be obtained while a patient is on the radiation treatment table.(A CT scan uses x-rays to produce detailed pictures of structures in the body.) In this study, cone beam CT scans will be obtained before individual radiation treatment sessions for head and neck cancer. The information gathered from these scans will be used by the researchers to look at patient movement as well as changes in the amount of normal and tumor tissue throughout the course of radiation therapy. The researchers will use this information to create hypothetical radiation treatment plans, which will be used as the basis for future research. The cone beam CT scan data will not be used to alter the actual radiation treatment of any of the patients enrolled on the study. In addition, tests of salivary output and swallowing and questionnaires about quality of life will be made to assess how the doses of radiation affect them.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages ≥18, both sexes, and all races will be included in this study. Pregnant females will be excluded. No other special classes of subjects (i.e., prisoners) will be entered.
* Patients must be diagnosed with biopsy-proven squamous cell carcinoma of the head and neck.
* Patients must be recommended treatment with definitive radiation therapy with concurrent chemotherapy, but without prior surgical resection of the primary tumor or lymph nodes
* Patients must be recommended a treatment course of at least 30 radiation fractions
* Patients must sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Michigan Hospital indicating that they are aware that undergoing cone beam CT of the head and neck is voluntary and has potential risks.

Exclusion Criteria:

* Patients must not have a history of prior radiation to the head or neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Eisbruch, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Hunter KU, Fernandes LL, Vineberg KA, McShan D, Antonuk AE, Cornwall C, Feng M, Schipper MJ, Balter JM, Eisbruch A. Parotid glands dose-effect relationships based on their actually delivered doses: implications for adaptive replanning in radiation therapy of head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):676-82. doi: 10.1016/j.ijrobp.2013.07.040. Epub 2013 Sep 10. PMID 24035328

RESULTS

PARTICIPANT FLOW:
Groups:
- Cone Beam CT: For the purposes of this study patients will get CT scans every day for the length of their radiation therapy (in order to assess if CT every day provides additional information compared with CT scans performed less frequently).
  Radiotherapy will be delivered according to current guidelines.
  Imaging will be performed every day before treatment for a total of approximately 35 cone beam CT scans over the 7 week course of therapy.
Period: Overall Study
Arm/Group | Cone Beam CT
Started | 23
Completed | 18
Not Completed | 5
Not completed — Completed Treatment Off Study | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Although 23 patients were enrolled, only 18 completed treatment.
Arm/Group | Cone Beam CT
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 57 [50 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Disease Site [Number; unit: participants] — Location of the disease at baseline.
  participants
    Base of Tongue | 9
    Tonsil | 9
T Stage [Number; unit: participants] — The T stage represents the size and stage of the primary tumor:
  TX: Primary tumor cannot be evaluated T0: No evidence of primary tumor Tis: Carcinoma in situ (CIS; abnormal cells are present but have not spread to neighboring tissue; although not cancer, CIS may become cancer and is sometimes called preinvasive cancer) T1, T2, T3, T4: Size and/or extent of the primary tumor (higher numbers represent more extensive disease)
  participants
    T1 | 2
    T2 | 10
    T3 | 5
    T4 | 1
N Stage [Number; unit: participants] — The N stage represents the amount of spread to nearby lymph nodes:
  NX: Regional lymph nodes cannot be evaluated N0: No regional lymph node involvement N1, N2, N3: Degree of regional lymph node involvement (number and location of lymph nodes)
  participants
    N0 | 1
    N1 | 0
    N2a | 1
    N2b | 10
    N2c | 4
    N3 | 2
Pre-Treatment Weight [Median (Full Range); unit: lb] | 203 [105 to 308]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Movement of Normal Tissue
Description: The primary outcome measure of this study is to characterize patient-specific target and normal tissue movement.
Time Frame: approximately 7 weeks
Reporting Status: Not Posted

2. Secondary Outcome: Improvement of Image Quality
Description: Use acquired data to further improve cone beam CT reconstruction techniques and image quality.
Time Frame: 36 months
Reporting Status: Not Posted

3. Secondary Outcome: The Median Delivered Dose of Radiation to the Parotid Gland
Time Frame: 7 weeks
Measure: Median (Full Range); unit: Gy
Arm/Group | Cone Beam CT
Number analyzed (Participants) | 18
Gy | 32.4 [23.2 to 63.2]

4. Primary Outcome: Correlation Coefficient for the Association Between Delivered Mean Parotid Dose and Salivary Flow Rate
Description: Spearman rank-based correlation coefficients were calculated for the association between saliva flow rate and the delivered mean parotid doses at several timepoints (Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months).
Time Frame: 24 months
Population: 36 parotid glands were evaluable from 18 patients at baseline, 34 parotid glands were evaluable at 3-6 months, 32 glands were evaluable at 12 months, 20 were evaluable at 18 months and 8 at 24 months.
Measure: Number; unit: correlation coefficient
Arm/Group | Cone Beam CT
Number analyzed (Participants) | 18
correlation coefficient
  Baseline | -0.26
  3 Months | -0.42
  6 Months | -0.57
  12 Months | -0.35
  18 Months | -0.42
  24 Months | -0.60

ADVERSE EVENTS:
Arm/Group | Cone Beam CT
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 9/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cone Beam CT (N=18)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cone Beam CT (N=18)
Chemoradiation Rash (Skin and subcutaneous tissue disorders) | 7 (12)
Radiation Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 8 (15)
xerostomia (Gastrointestinal disorders) | 9 (30)
Dysphagia (Gastrointestinal disorders) | 9 (21)
Esophagitis (Gastrointestinal disorders) | 8 (17)
Gastrointestinal Other (Gastrointestinal disorders) | 2 (7)
Mucositis/Stomatitis (upon exam) (Investigations) | 9 (25)
Mucositis/Stomatitis (symptomatic) (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Salivary Gland Changes (Gastrointestinal disorders) | 7 (22)
Dysgeusia (Gastrointestinal disorders) | 9 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes